CLINICAL TRIAL: NCT00845533
Title: Pharmacokinetics of Dihydroartemisinin-Piperaquine in the Treatment of Uncomplicated Malaria in Children in Burkina Faso
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Holley-Cotec Pharmaceuticals Co., LTD. (Unknown); Mahidol University (Other)
Responsible Party: Principal Investigator, Sunil Parikh, Assistant Professor, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H40380-31179-01
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Uncomplicated Malaria

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine

SUMMARY:
This will be an open-label trial in Burkina Faso assessing the pharmacokinetics of the antimalarial combination of dihydroartemisinin/piperaquine (DP, Duocotexcin) in children. Dihydroartemisinin-piperaquine is a promising candidate for first-line therapy of malaria. We hypothesize that the disposition and pharmacokinetics of DP will be altered in children, and this will alter the efficacy and/or toxicity of DP. We will test this hypothesis in this open-label trial in Burkina Faso. The target population includes residents, aged 6 months to 10 years in Bobo-Dioulasso. Children who present to the study clinics with symptoms suggestive of malaria will be screened with a thick blood smear. Subjects who meet selection criteria of treatment efficacy will be treated and followed up for 42 days. Pharmacokinetic sampling for DP will occur on selected follow-up days.

ELIGIBILITY:
Inclusion Criteria:

1. Positive screening thick blood smear
2. Fever (> 37.5ºC axillary) or history of fever in the previous 24 hours
3. Age ≥ 6 months to 10 years
4. Weight > 5 kg
5. Absence of any history of serious side effects to study medications
6. No evidence of a concomitant febrile illness in addition to malaria
7. No history of antimalarial use in the previous two weeks
8. P. falciparum mono-infection
9. Parasite density 2000-200,000/ul
10. Provision of informed consent and ability to participate in 42-day follow-up

Exclusion Criteria:

1. Danger signs or evidence of severe malaria
2. Hemoglobin levels < 5.0 gm/dL

Ages: 6 Months to 10 Years | Sex: All
Age Groups: Child
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Parikh, M.D., M.P.H., Principal Investigator — University of California, San Francisco; Philip J Rosenthal, M.D., Principal Investigator — University of California, San Francsico; Jean-Bosco Ouedraogo, M.D., PhD, Principal Investigator — Institut de Receherche en Sciences de la Sante Bobo-Dioulasso